CLINICAL TRIAL: NCT05151016
Title: A Multicenter Randomized Clinical Trial of Mifepristone Versus GnRHa for the Treatment of Adenomyosis
Brief Title: Long-term Use of Mifepristone in the Treatment of Adenomyosis
Acronym: LUOMITTOA
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Ningbo Women & Children's Hospital (Other); Jiaxing Maternity and Child Health Care Hospital (Other); The Affiliated Hospital of Medical School, Ningbo University (Unknown); Qilu Hospital of Shandong University (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210229
Record Dates: First submitted 2021-10-07; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Adenomyosis; Mifepristone
MeSH Terms: conditions — Adenomyosis | interventions — Mifepristone; Triptorelin Pamoate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mifepristone (Experimental): mifepristone tablets，10mg，One tablet daily, oral treatment
  Interventions: Drug: mifepristone
- Triptorelin Acetate (Active Comparator): dafinil, 3.75 mg, first injection on the third day of menstruation, followed by intramuscular injection every 28 days for 24 weeks.
  Interventions: Drug: Triptorelin Acetate

INTERVENTIONS:
Drug: mifepristone — Mifepristone tablets, 10mg, 1 tablet daily, taken orally (beginning on the third day of Menstruation) for 24 weeks
  Arms: mifepristone
Drug: Triptorelin Acetate — dafinil, 3.75 mg, first injection on the third day of menstruation, followed by intramuscular injection every 28 days for 24 weeks.
  Arms: Triptorelin Acetate

SUMMARY:
The design was a prospective, randomized, positive-control, parallel-group, multicenter clinical trial. The study included a randomized, parallel-group treatment for 24 weeks in 140 subjects from eight hospitals in seven cities across the country who were diagnosed with Adenomyosis and associated symptoms (dysmenorrhea, with or without heavy menstrual flow) , the subjects were randomly assigned to the following two groups:

1. Study Group: mifepristone tablets, 10 mg, 1 tablet daily, taken orally (beginning on the third day of Menstruation) for 24 weeks;
2. Control Group: dafinil (Triptorelin Acetate) , 3.75 mg, first injection on the third day of menstruation, followed by intramuscular injection every 28 days for 24 weeks.

ELIGIBILITY:
Inclusion criteria.

* Female, over 18 years old and not menopausal, agree to tripriline acetate and mifepristone treatment and informed consent
* Patients were diagnosed as adenomyosis by postoperative pathology, or those who did not undergo surgery but were diagnosed by auxiliary examination, such as ultrasonography and MRI.
* Dysmenorrhea with or Without Menorrhagia
* Requiring preservation of the uterus or fertility
* No other hormonal treatment for Adenomyosis was received in the three months prior to treatment
* Normal or non-clinically significant cervical cytology results (6 months before the screening period)

Exclusion criteria.

* Pelvic pain and vaginal bleeding of unknown or non-Adenomyosis causes
* Benign Lesions such as endometrial polyp, submucous Myoma or suspicious malignant tumors were diagnosed by ultrasonography
* Receiving other hormone drugs for Adenomyosis
* Use other drugs that interact with tripriline acetate and mifepristone, and can not be stopped
* Patients with severe heart, liver, kidney disease and Adrenal insufficiency; drug allergy or allergic constitution
* Participated in other clinical trials within 3 months, and other factors considered unsuitable for the trial
* Pregnant, lactating women and those who prepare for childbirth during the treatment or within six months after treatment
* Postmenopausal women.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pain on the Visual Analogue Scale (VAS) at week 24 | Baseline and Week 24
  The VAS is the most commonly used instrument assessing pain in clinical practice. It reflects the patient's subjective perception of pain. Possible scores range from 0 (no pain) to 10 (worst possible pain). The last observation carry forward was used for missing data.
  Change=(Week 24 Score - Baseline Score)

SECONDARY OUTCOMES:
Pictorial blood loss assessment chart（PBAC） | Baseline and week 24
  Recording the use of tampons and sanitary towels by placing a tally mark under the day next to the box. Record clots by indicating whether they are the size of a 1p or 50pcoin in the clots/ flooding row under the relevant day. E.g. under day1 you may say 50p*1 and 1p*3. Record any incidences of flooding by placing a tally mark in the clots/ flooding row under the relevant day. A lightly stained towel (pic 1) will score 1 point, a moderately stained towel (pic 2) 5 points, a towel which is saturated with blood(pic 3) will score 20 points. A lightly stained tampon (pic 4) will score 1 point, a moderately stained tampon (pic 5) 5 points and a tampon that is fully saturated will score 10 points. A clot the size of 1p scores 1 point, a 50p sized clot scores 5 pointsand flooding also scores 5 points. Finally, total up the scores. A score of100 or greater may indicate a heavy period.
  Change=Week 24 Score - Baseline Score
Change from baseline in uterine size at week 24 | Baseline and week 24
  Uterine size usually reflects the size of the adenomyosis lesion, and is measured in cubic centimeters.
  Change=(Week 24 Uterine Size - Baseline Uterine Size)*0.5236
Change from baseline in hemoglobin at week 24 | Baseline and week 24
  Hemoglobin, measured in grams per liter, reflects a patient's level of menstrual blood loss.
  Change=(Week 24 Hemoglobin Content - Baseline Hemoglobin Content)
Change from baseline in CA125 at week 24 | Baseline and week 24
  CA125 is measured in micrograms per liter. Change=(Week 24 Hemoglobin Content - Baseline Hemoglobin Content)

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital of Zhejiang Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided